CLINICAL TRIAL: NCT06640179
Title: Prevention of Weight Gain and Impaired Glucose Metabolism Post Kidney Transplantation: A Pilot and Feasibility Study
Brief Title: Feasibility and Plausible Effectiveness of a Lifestyle Intervention in Kidney Transplant Recipients (HEAL)
Acronym: HEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John M. Jakicic, PhD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY001680081; R01DK137986-01 (NIH)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant; Overweight or Obese Adults; Glucose Control
Keywords: kidney transplant; overweight; obesity; glucose control; weight control
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Care (Active Comparator): Standard Care Intervention will continue to receive their regular standard clinical care during the 6-month intervention period of this study and will also receive brief conducts (<10 minutes) from the research staff at weeks 6, 12, and 18.
  Interventions: Other: Standard medical care; Behavioral: Monitoring Contacts
- Standard Medical Care plus Lifestyle Intervention (Experimental): Standard Medical Care plus Lifestyle Intervention will continue to receive their regular standard clinical care and a behavioral intervention focused on dietary modification and physical activity for body weight regulation.
  Interventions: Other: Standard medical care; Behavioral: Behavioral Sessions; Behavioral: Diet; Behavioral: Physical Activity

INTERVENTIONS:
Other: Standard medical care — Standard Care Intervention will continue to receive their regular standard clinical care during the 6-month intervention period of this study.
Behavioral: Monitoring Contacts — Participants will receive brief conducts (<10 minutes) remotely (telephone or video platform) with the research staff at weeks 6, 12, and 18.
  Arms: Standard Medical Care
Behavioral: Behavioral Sessions — Participants will be provided weekly individual behavioral sessions during the 6-month intervention to assist in supporting recommended changes in energy intake (diet) and physical activity.
  Arms: Standard Medical Care plus Lifestyle Intervention
Behavioral: Diet — An energy balanced diet to meet energy needs that will allow for weight maintenance will be prescribed. This will be estimated using the Mifflin-St. Joer equation to estimate resting metabolic rate and for most participants we anticipate using a physical activity correction of 1.3 to account for energy needs for physical activity. This will provide the initial estimate of energy intake needs to maintain weight stability; however, the prescribed level of energy intake will be adjusted at 4-week intervals across the intervention based on the observed changes in weight, eating behaviors, and physical activity patterns in an effort to prevent excessive weight gain. Within the context of this level of energy intake, we will prescribe a diet that is consistent with the dietary recommendations of the National Kidney Foundation.
  Arms: Standard Medical Care plus Lifestyle Intervention
Behavioral: Physical Activity — Physical activity will be recommended in the form of aerobic types of activity such as brisk walking and will progress in 4-week intervals from an initial amount of 50 minutes per week to 150 minutes per week across the initial 6 months of the intervention. Moderate intensity will be prescribed, and will be anchored using RPE (rating of perceived exertion) to allow intensity to be self-regulated according to the participant's capacity. Physical activity will be prescribed in the form of walking; however, the participant will be permitted to engage in other forms of physical activity that meet the recommended dose and intensity.
  Arms: Standard Medical Care plus Lifestyle Intervention

SUMMARY:
The goal of this clinical trial is to learn whether if it is feasible to implement a study of patients receiving kidney transplantation, to learn if these patients will complete selective outcomes measurements, and to examine if a lifestyle intervention may assist with preventing weight gain compared to standard medical care. The main questions it aims to answer are:

* Is it feasible to recruit and retain patients who have undergone kidney transplantation into a study to compare standard medical care to standard medical care plus a lifestyle intervention focused on prevention of weight gain?
* Will participants engage in the interventions and be compliant to the components of the interventions?
* Will there be any difference between the interventions between the interventions for the occurrence of adverse events specific to kidney transplantation?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on preventing weight gain compared to standard medical care alone?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on body composition compared to standard medical care alone?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on fasting glucose compared to standard medical care alone?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on fasting insulin compared to standard medical care alone?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on insulin sensitivity compared to standard medical care alone?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on physical function compared to standard medical care alone?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on health-related quality of life compared to standard medical care alone?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on changes in dietary intake compared to standard medical care alone?
* Will there be initial effectiveness for the standard medical care plus a lifestyle intervention to have a better effect on physical activity and sedentary behavior compared to standard medical care alone?

Participants will:

* Participants will continue with their standard medical care following kidney transplantation.
* Participants only receiving standard medical care will also complete brief monitoring visits at week 6, 12, and 18.
* Participants receiving the lifestyle intervention will attend weekly intervention sessions and will be recommended to modify their diet and physical activity behaviors in an effort to prevent weight gain.
* Participants will complete outcome measurements as the start of the study and again after 6 months in the study.
* After 6 months in the study, participants will also complete a brief intervention and answer other questions about their experience in the study.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a kidney transplant within the prior 3-5 months, with the transplant received from a deceased donor or living donor. NOTE: The patient will be eligible for randomization at 3 months following the kidney transplant, or at a subsequent time once clearance from the kidney transplant physician is given, provided that the time does not exceed 5 months following the kidney transplant.
* Both males and females of all race/ethnic groups are eligible for participation in this study.
* >=18 years of age.
* Body mass index (BMI) >22 kg/m2. There is no maximal BMI provided that the weight does not exceed the weight allowance of the dual-energy x-ray absorptiometer (DXA) that is used to assess body composition (maximal weight for the DXA is 350 pounds).
* Ability to provide informed consent prior to participation in this study.
* Ability to provide clearance from their kidney transplant physician to engage in the diet and physical activity components of the proposed intervention and to safely complete the proposed outcome measures.
* Ability to walk for exercise.

Exclusion Criteria:

* Females who are pregnant, breastfeeding, or reporting a planned pregnancy during the study period. Female participants of childbearing age who are not currently taking contraceptive medication, are not post-menopausal, or have not been surgically sterilized will need to agree to use a double barrier method of contraception.
* History of bariatric surgery.
* Currently prescribed an anti-obesity medication.
* Report current medical condition or treatment for a medical condition that could affect body weight. These may include the following: diabetes mellitus; hyperthyroidism; inadequately controlled hypothyroidism; chronic liver disease; cancer; gastrointestinal disorders including ulcerative colitis, Crohn's disease, or malabsorption syndromes; etc.
* Current congestive heart failure, angina, uncontrolled arrhythmia, symptoms indicative of an increased acute risk for a cardiovascular event, prior myocardial infarction, coronary artery bypass grafting or angioplasty, conditions requiring chronic anticoagulation (i.e., recent or recurrent DVT).
* Resting systolic blood pressure of >=160 mmHg or resting diastolic blood pressure of >=100 mmHg or not on a stable medical treatment to control hypertension (stable dose is defined as the same dose and type of medication for a period of at least 6 months).
* Eating disorders that would contraindicate modifying eating or physical activity behaviors.
* Alcohol or substance abuse.
* Currently treated for psychological issues (i.e., depression, bipolar disorder, etc.) that is accompanied by the following: 1) not on a stable dose of medications for treatment within the previous 12 months, or 2) hospitalized for depression within the previous 5 years.
* Report plans to relocate to a location not accessible to the study site or having employment, personal, or travel commitments that prohibit attendance at scheduled intervention sessions or assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 0 and 6 months
  Body weight will be assessed in duplicate using a calibrated digital scale to the nearest 0.1 kg.

SECONDARY OUTCOMES:
Body Mass Index | 0 and 6 months
  Measurements of weight and height will be used to compute BMI (kg/m2).
Percent body fat | 0 and 6 months
  Percent body fat will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Body Fat Mass | 0 and 6 months
  Body fat mass (kg) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Lean Body Mass | 0 and 6 months
  Lean body mass (kg) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Bone mineral content | 0 and 6 months
  Bone mineral content (grams) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Waist Circumference | 0 and 6 months
  Circumference measures of the waist taken horizontally at both the iliac crest and the umbilicus will be performed.
Hip Circumference | 0 and 6 months
  Circumference measures of the hip taken horizontally at widest portion of the buttocks will be performed.
Resting blood pressure | 0 and 6 months
  Resting blood pressure will be measured in duplicate following a 5-minute seated rest period using an automated measuring system.
Resting heart rate | 0 and 6 months
  Resting heart rate will be measured following a 5-minute seated rest period using an automated measuring system.
Physical Function | 0 and 6 months
  Physical function will be measured with a 400-meter walk test. The score will be the duration of time (minutes) it takes to complete the 400 meters.
Fasting glucose | 0 and 6 months
  Fasting glucose will be measured from a blood sample collected after at least an 8-hour fasting period.
Fasting Insulin | 0 and 6 months
  Fasting insulin will be measured from a blood sample collected after at least an 8-hour fasting period.
Insulin Resistance | 0 and 6 months
  HOMA-IR will be used as a measure of Insulin resistance, which is computed from measures of fasting glucose and fasting insulin.
Kidney function | 0 and 6 months
  Kidney function will be measured using glomerular filtration rate (GFR) measured from a blood sample after at least 8 hours of fasting.
Physical activity | 0 and 6 months
  Physical activity will be assessed with the Paffenbarger questionnaire that queries on walking, flights of stairs climbed, and other sport, recreational, or leisure physic activity. Physical activity is represented by the total minutes of activity per week and estimated kilocalories of physical activity per week.
Physical Activity | 0 and 6 months
  Physical activity is measured by the Global Physical Activity Questionnaire (GPAQ). This assesses time spent in recreational, occupational, household, and transportation physical activities and is represented as minutes per week.
Sedentary behavior | 0 and 6 months
  Sedentary behavior is measured using an 8-item survey that is completed for weekdays and weekend days. Time spent in sedentary behavior is reported.
Energy Intake (Dietary Intake) | 0 and 6 months
  Energy Intake (Dietary Intake) expressed as kilocalories eaten per day (kcal/day) will be measured using the Diet History Questionnaire (DHQ) developed by NCI. A higher score represents more calories eaten.
Weight Loss Strategies | 0 and 6 months
  Weight Loss Strategies will be measured using the Weight Control Strategies Scale that includes 30 items. Each item is scored on a 0-4 scale and the scores across the 30 items are summed to provide an overall score, with a range for the total score being 0 to 120. A higher score is more favorable and represents engaging in more weight control strategies.
Weight Loss Strategies | 0 and 6 months
  Weight Loss Strategies will be measured using the Eating Behavior Inventory that includes 26 items with each measured on a 5-point scale. The score from each item is summed for a total score, with the being 26-130. A higher score represents engaging in more appropriate weight loss strategies.
Health-Related Quality of Life | 0 and 6 months
  Health-Related Quality of Life will be measured with a 36-item questionnaire (RAND 36-Item Health Survey) that includes 8 subscales of vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health or emotional wellbeing. All items are scored so that a high score defines a more favorable health state. The range of the final score for each subscale is 0-100.
Adverse and Serious Adverse Events | 0 and 6 months and at other times when reported by the participant
  Participants will be queried using a survey developed specifically for this study will be used to assess for adverse events and serious adverse events.

OTHER OUTCOMES:
Medication History | 0 and 6 months
  A questionnaire developed specifically for this study will be used to assessment medication history. The data collected include the type of medication, dose of medication, and frequency that the medication is taken, and what condition the medication is indicated to treat.
Lifestyle and Health History | 0 months (prior to randomization)
  A questionnaire developed specifically for this study that is conducted as an interview will be used to assess lifestyle and health factors to describe the sample for this study. The score is either "yes" or "no" identifying the presences of a lifestyle or health factor.
Post-Intervention Qualitative Interview | 6 months
  Each participant will undergo a qualitative interview in a face-to-face format to allow the investigators to better understand strengths, weaknesses, and barriers that will allow for further intervention refinement prior to proceeding a larger study.
Post-Intervention Qualitative Questionnaire | 6 months
  Each participant will complete a questionnaire to allow the investigators to better understand strengths, weaknesses, and barriers that will allow for further intervention refinement prior to proceeding a larger study.

CONTACTS AND LOCATIONS:
Overall Officials: John M. Jakicic, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The summary data for each of the study outcomes and other additional demographic characteristics will be made available. The Study Protocol (which includes the statistical analysis plan), Manual of Procedures, Data Collection Forms, and a Data Dictionary to explain the data variables will be provided.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available no later than the time of an associated publication of study outcomes or at the end of the performance period, whichever comes first. The data provided to the repository will be available indefinitely while that repository continues to exist.
Access Criteria: The information included with the IPD will be made available to appropriate individuals only after the requester confirms their willingness to comply with an appropriate "Data Use Agreement" that complies with NIH policies, the policies of the institution where the study has been conducted, and the elements of informed consent.